CLINICAL TRIAL: NCT01063192
Title: A Phase II Randomized Study of Induction Chemotherapy Followed by Concurrent Chemo-radiotherapy in Locally Advanced Pancreatic Cancer
Brief Title: A Study of Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: National Health Research Instiutes, Taiwan, National Institute of Cancer Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2209
Record Dates: First submitted 2009-11-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Gemcitabine; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine (Active Comparator): Arm 1: Gemcitabine alone
  Interventions: Drug: Gemcitabine
- GOFL (Active Comparator): Arm 2: GOFL (Gem 800mg/m2 80min, Oxa 85mg/m2 2hr, 5FU 3000mg/m2, LV 150mg/m2 iv 48hr)
  Interventions: Drug: Gemcitabine, Oxaliplatin, 5-Fluorouracil, Leucovorin (GOFL)

INTERVENTIONS:
Drug: Gemcitabine — Arm 1: Gemcitabine alone on D1,8,15 every 28 days for 3 cycles
  Arms: Gemcitabine
Drug: Gemcitabine, Oxaliplatin, 5-Fluorouracil, Leucovorin (GOFL) — Arm 2: GOFL on D1, 15 every 28 days for 3 cycles(Gem 800mg/m2 80min, Oxa 85mg/m2 2hr, 5FU 3000mg/m2, LV 150mg/m2 iv 48hr)
  Arms: GOFL

SUMMARY:
The primary end point is to evaluate the time to progression after gemcitabine alone versus Gemcitabine-based combination induction chemotherapy followed by concurrent chemoradiotherapy in locally advanced pancreatic cancer.

The secondary end points are to evaluate the disease control rate, overall survival time, toxicity profile and compliance after induction chemotherapy and concurrent chemoradiotherapy as well as the disease control rate after inductional chemotherapy alone in locally advanced pancreatic cancer. Translational research including pharmacogenomic study and biomarker study will also be done concomitantly.

DETAILED DESCRIPTION:
Patients should be randomized to two study arms stratified by resectability status (borderline resectable and unresectable) after enrollment. Eligible patients will be randomly assigned on a 1:1 basis to either of two study groups, using a central randomization procedure with stratification according to NCCN criteria of resectability.

After randomization, induction chemotherapy (ICT) will be administered for 3 cycles ( 3 months). Patients who have radiological evidence of distant dissemination will be shifted to salvage chemotherapy. Patients who have responsive, stable disease as well as those with localized progressive disease after ICT will receive concurrent chemoradiotherapy (CCRT) 3-4 weeks after the last dose of ICT. Surgical evaluation will be performed 4-6 weeks after the completion of CCRT. Patients who have respectable disease will undergo surgical resection. Postoperative adjuvant chemotherapy for 3 cycles ( 3 months) will be given for those who are considered to have curative resection. Patients who still have unresectable disease or non-curative resection will receive systemic chemotherapy till disease progression or unacceptable toxicity.

For Arm 1, ICT with gemcitabine ( fixed rate of 10mg/m2/min, 1000mg/m2 on day 1,8,15 every 28 days/cycle) will be administered on a 3-week-on-one-week-off weekly basis. For Arm 2, ICT with GOFL ( 800mg/m2 gemcitabine at a fixed rate of 10mg/m2/min followed by a 2-hour oxaliplatin 85mg/m2 and then a 48-hour 3000mg/m2 5-FU and 150 mg/m2 leucovorin on day 1 and 15 every 28 days/cycle) will be given biweekly.

After three 3 cycles of ICT, patients without distant metastasis will be given CCRT with gemcitabine 400mg/m2 2 hrs before RT on day1,8,15,22,29,36. Radiation will be given 180cGy per day, 5 days a week for 28 fractions to totally 5040cGy.

If complete surgical resection is feasible, optimal surgery will be performed 4-6 weeks after CCRT. If complete surgical resection is impossible, biopsy with or without bypass surgery may be performed. Patients who have curative surgical resection will receive additional 6 cycles ( 6 months) of adjuvant chemotherapy ( Arm1, gemcitabine alone; Arm 2, GOFL) within 4 weeks after surgery and then followed up until tumor progression. Patients who are not feasible for curative resection, will receive continued chemotherapy (Arm1, gemcitabine alone; Arm2, GOFL) 3-4 weeks after CCRT complete. The regimen will continue till disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the exocrine pancreas.
2. Patients must have locally advanced pancreatic cancer (LAPC).
3. Patients must have LAPC evaluated by radiologist and/or surgeon according to either abdominal CT or MRI, or intra-operative findings.
4. Patients must have measurable disease.
5. Age >20 years.
6. ECOG performance scale of 0-2.
7. Patients must have normal organ and marrow function.
8. Patients who present with jaundice, temporary or permanent internal / external drainage before enrollment will be allowed.
9. The effects of study agents on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with distant metastases are not eligible.
2. Patients may not be receiving any other investigational agents.
3. Patients who have had prior chemotherapy or radiotherapy are not eligible.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents used in the study.
5. Patients who have above grade II peripheral neuropathy.
6. Patients who had non-curable second primary malignancy.
7. Uncontrolled intercurrent illness including.
8. Pregnant women are excluded from this study because the study agents has the potential for teratogenic or abortifacient effects.
9. Those who are immuno-compromised or receiving immuno-suppressive therapy are excluded from the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to evaluate the time to progression after gemcitabine alone versus Gemcitabine-based combination induction chemotherapy followed by concurrent chemoradiotherapy in locally advanced pancreatic cancer. | 6 months

SECONDARY OUTCOMES:
The secondary end points are to evaluate the disease control rate, overall survival time, toxicity profile and compliance after induction chemotherapy and concurrent chemoradiotherapy . | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Wen Lin, M.D, Study Chair — National Cheng-Kung University Hospital; Yen-Shen Shen, M.D., Principal Investigator — National Cheng-Kung University Hospital; Chiun Hsu, Ph.D., Principal Investigator — National Taiwan University Hospital